CLINICAL TRIAL: NCT01858116
Title: An Exploratory Study to Evaluate [68Ga]ABY-025 for PET Imaging of HER2 Expression in Subjects With Metastatic Breast Cancer
Brief Title: PET Study of Breast Cancer Patients Using [68Ga]ABY-025
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomedical Radiation Sciences (Other)
Collaborators: Swedish Cancer Society (Other); Affibody (Industry)
Responsible Party: Principal Investigator, Dr. Henrik Lindman, Oncology, Chief Physician, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABY-025-MI105; 2012-005228-14 (EudraCT Number)
Record Dates: First submitted 2013-04-12; First posted 2013-05-21 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 68Ga-ABY-025

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [68Ga]ABY-025 (Experimental)
  Interventions: Drug: [68Ga]ABY-025

INTERVENTIONS:
Drug: [68Ga]ABY-025 — Intravenous injection followed by PET imaging

SUMMARY:
The study will evaluate [68Ga]ABY-025 for PET imaging of HER2 expression in subjects with HER2-positive or HER2-negative breast cancer.

DETAILED DESCRIPTION:
Open-labeled, exploratory, single center study.

1. Group 1 (dose-finding) Six subjects with HER2-positive primary tumor status and four subjects with HER2-negative status. [68Ga]ABY-025 PET with low dose (100 μg) of ABY-025 peptide is performed, followed by a repeated PET within three weeks using high dose (500 μg) ABY-025 peptide (radioactivity maximum 500 MBq). A third [68Ga]ABY-025 PET will be performed in the HER2-positive subgroup only, when signs of progressive disease are found at routine clinical evaluation or else latest after 12 months regardless of disease status, then using the ABY-025 peptide dose previously determined to be preferable.
2. Group 2 Ten subjects with HER2-positive primary tumor status. [68Ga]ABY-025 PET is performed using the ABY-025 peptide dose determined to be preferable during the dose-finding part of the study, followed by a second [68Ga]ABY-025 PET investigation at signs of progressive disease or else latest after 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Diagnosis of invasive breast cancer with metastases
3. Availability of results from HER2 status previously determined on material from the primary tumor, either

   1. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or
   2. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+ or else; if 2+ then FISH negative
4. Volumetrically quantifiable metastasis lesions on CT or MRI, with at least one lesion >= 10 mm in smallest diameter and suitable for biopsy
5. ECOG performance status of =< 2
6. Life expectancy of at least 12 weeks
7. Hematological, liver and renal function test results within the following limits:

   White blood cell count: > 2.0 x 10^9/L Haemoglobin: > 80 g/L Platelets: > 50.0 x 10^9/L ALT, ALP, AST: =< 5.0 times Upper Limit of Normal Bilirubin =< 2.0 times Upper Limit of Normal Serum creatinine: Within Normal Limits or else normal clearance
8. A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all female patients of childbearing potential, who must use a medically acceptable form of contraception from study start until at least 30 days after study termination
9. Subject is able to participate in the diagnostic investigations to be performed in the study
10. Informed consent

Exclusion Criteria:

1. Manifest second, non-breast malignancy
2. Known HIV positive or chronically active hepatitis B or C
3. Administration of other investigational medicinal product within 30 days of screening
4. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's "Common Terminology Criteria for Adverse Events v4.0 [CTCAE]"
5. Other ongoing severe disease that may influence the patient's ability to participate in the study
6. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
PET image analysis: Standardized Uptake Value (SUV) and uptake kinetics of [68Ga]ABY-025 in breast cancer lesions and normal tissues | Day 0

SECONDARY OUTCOMES:
SUV in metastases where biopsy results with HER2 status by IHC/FISH are available | Day 0
SUV for each measured lesion, and appearance or disappearance of lesions, after progression or 9-12 months therapy | Up to 1 year
SUV for each measured lesion and number of detectable lesions, obtained with a low (100 μg) or high (500 μg) injected amount of ABY-025 peptide in the same subject | Day 0 & 1-3 weeks
SUVs for all measured lesions obtained with a low (100 μg) or high (500 μg) injected where biopsy results with HER2 status by IHC and FISH are available | Day 0
Incidence and severity of adverse events | Day 0 to 42
Anti-Drug Antibody assay at 3 and 6 weeks | Day 0 to 42
Blood radioactivity kinetics and dosimetry of [68Ga]ABY-025 | Day 0
Uptake of [68Ga]ABY-025 coinciding with metastatic lesions visible on [18F]FDG PET and focal uptake in regions without pathological findings on [18F]FDG PET | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Lindman, MD, PhD, Principal Investigator — Uppsala University Hospital, Department of Oncology
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden